CLINICAL TRIAL: NCT04633369
Title: The Role of the Microbiome and Host Physiology in Personalized Human Response to Dietary Fibers Intake During Intermediate Fasting
Brief Title: The Role of the Microbiome in the Response to Dietary Fibers Intake During Intermediate Fasting
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weizmann Institute of Science (Other)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MHO-0488-20
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-02

CONDITIONS: Dietary Fibers; Intermediate Fasting
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fructo-oligosaccharide (Experimental): Fructo-oligosaccharide 20g
  Interventions: Dietary Supplement: dietary fibers
- Arabinogalactan (Experimental): Arabinogalactan 12g
  Interventions: Dietary Supplement: dietary fibers
- Glucomannan (Experimental): Glucomannan 4g
  Interventions: Dietary Supplement: dietary fibers

INTERVENTIONS:
Dietary Supplement: dietary fibers — during days 13-22 the participants will consume the dietary fiber according to their randomization and continue fasting. Participants will be asked to collect stool and oral samples 4 times during this period.

SUMMARY:
Dietary fibers are generally not degraded by the endogenous digestive enzymes, but rather by the complex ensemble of microorganisms that reside in the human gut [1]. This ensemble, collectively known as the human gut microbiome, plays a key role in breaking down, fermenting, and ultimately converting such dietary fibers into a variety of beneficial metabolites, including most notably, short chain fatty acids (SCFA). These end products of fibers' fermentation affect host metabolism, immunity, and physiology, and have been implicated in multiple diseases including obesity, metabolic syndrome, diabetes, and cardiovascular diseases.

Intermediate fasting, and in particular circadian intermediate fasting (i.e. 16 hours of fasting followed by 8 hours of allowed eating), has been shown to have positive associations with multiple health conditions as obesity, diabetes mellitus, cardiovascular disease, cancers, and neurologic disorders In this study, we will try to answer open questions utilizing the long fasting period during the day to investigate the isolated effect of dietary fiber consumption, uncovering the degradation effect, but not the bulking effect, on the microbiome and the host physiology, and in particular its glucose response.

DETAILED DESCRIPTION:
During the 22 days of the study, participants will wear a continuous glucose monitor, fill a daily food diary, and collect stool and oral samples which will be used for microbiota profiling. Participants will be asked to carry out an intermediate fasting regime, which will include: 16 straight hours of fasting followed by 8 hours which the participants will be allowed to eat. Drinking water is allowed throughout the fasting hours.

The groups will consume 4, 12, 20 grams of the dietary fiber per day, according to the group they were assigned to, while not exceeding the total fiber consumption of 50 grams per day, which is considered a high-fiber diet.

ELIGIBILITY:
Inclusion Criteria:

Male and Female BMI<28 Age - 18-70

Exclusion Criteria:

Consumption of antibiotics 3 months prior to the first day of the experiment. Consumption of probiotic or dietary fibers supplements 1 month prior to the first day of the experiment.

Practiced in intermediate fasting 1 month prior to the first day of the experiment.

Diagnosis with type 1 or type 2 diabetes. Pregnancy, breastfeeding, or fertility treatments in the last 6 months. Chronic disease (e.g. AIDS, Cushing syndrome, CKD, acromegaly, hyperthyroidism hepatitis, fibromyalgia, etc.).

Cancer and recent anticancer treatment. Psychiatric disorders. Coagulation disorders. IBD (inflammatory bowel diseases). IBS (Irritable bowel syndrome). Alcohol abuse, more than 2 drinks per day for males, and more than one drink for females.

Substance abuse. BMI>28. Daily dietary intake higher than 25 grams per day. History of abdominal surgeries (including Bariatric surgery). Mentally incompetent or lack of judgment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
microbiome | 1 year
  stool and oral samples
glycemic response of different dietary fibers | 1 year
  Continuous glucose monitoring (CGM)

CONTACTS AND LOCATIONS:
Overall Officials: Eran Elinav, Prof, Principal Investigator — Weizmann Institute of Science
Locations (1):
- Weizmann institute of science, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: No